CLINICAL TRIAL: NCT00411619
Title: Everolimus (RAD001)Therapy of Giant Cell Astrocytomas in Patients With Tuberous Sclerosis Complex
Brief Title: Everolimus (RAD001) Therapy of Giant Cell Astrocytoma in Patients With Tuberous Sclerosis Complex
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCHMC IRB# 06-07-50
Record Dates: First submitted 2006-12-12; First posted 2006-12-14 (Estimated); Results first posted 2014-10-20 (Estimated); Last update posted 2014-10-20 (Estimated); Status verified 2014-10

CONDITIONS: Tuberous Sclerosis; Subependymal Giant Cell Astrocytoma
Keywords: Tuberous Sclerosis Complex (TSC); Subendymal Giant Cell Astrocytomas (SEGA'S); Mammalian Target of Rapamycin (mTOR); Everolimus (RAD001); Tuberous Sclerosis with Subependymal Giant Cell Astrocytomas
MeSH Terms: conditions — Tuberous Sclerosis; Astrocytoma; Hereditary Sensory and Autonomic Neuropathies | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Everolimus (Experimental): As this was a non-randomized, open-label, single arm study, all patients in the study received treatment with everolilmus
  Interventions: Drug: Everolimus

INTERVENTIONS:
Drug: Everolimus — Initial everolimus dosage will be 3 mg/m2/d taken daily or every other day, with titration to achieve a trough serum level of 5-15 ng/ml. Patients unable to tolerate levels in this range will have doses held or reduced 25% to achieve trough serum levels of 5-10 ng/ml. If trough serum level of 5-15 ng/ml is not achieved at a dosage of 3 mg/m2/d, then dosage escalation by 25% will be undertaken as tolerated. Everolimus will be similarly adjusted during the extension phase. If a subject misses more than 10 consecutive everolimus doses, additional days of everolimus treatment will be added so total duration of treatment is 6 months. If this occurs, dates of subsequent study events will be adjusted according to number of missed doses. This process will also be followed in the extension phase.
  Other Names: RAD001

SUMMARY:
The purpose of the study is to evaluate the safety and potential side effects of everolimus (an experimental drug) on a person with Tuberous Sclerosis Complex who also has been diagnosed with a brain tumor (astrocytoma)

The hypothesis is that the drug will cause the tumor size to decrease, and may have beneficial activity separate from effects on tumors in patients.

DETAILED DESCRIPTION:
Tuberous Sclerosis Complex (TSC)is a genetic disorder with a birth incidence of approximately one in six thousand. Five to twenty percent of patients with TSC will develop astrocytoma, a slowly progressive tumor. They grow and cause damage to surrounding brain tissue, blockage of spinal fluid (hydrocephalus), blindness, trouble walking, seizures, and brain damage. If untreated, they can be fatal. Standard treatment involves surgery to remove the tumor; however surgery may itself cause brain damage, bleeding, or infection, as well as other complications. Studies have shown that everolimus suppresses the chemicals that cause tumors to grow in tuberous sclerosis, and may cause them to shrink.

The primary objective of this study is to find out the effects of everolimus on astrocytomas in a six month trial in patients with Tuberous Sclerosis who have been diagnosed with an astrocytoma

ELIGIBILITY:
Inclusion Criteria:

* Age three years and older
* If female and of child bearing potential, documentation of negative pregnancy test prior to enrollment. In the extension phase, all females of child bearing potential will be required to take monthly home pregnancy tests and record results on a provided diary card.
* Clinically definite diagnosis of tuberous sclerosis (modified Gomez criteria or positive genetic test)
* Presence of giant cell astrocytoma as defined by imaging characteristics and serial increase in size of lesion on 2 or more MRI scans
* Adequate renal function (creatinine < 1.5 mg/dl)

Exclusion Criteria:

* Serious intercurrent medical illness or other uncontrolled medical disease which could compromise participation in the study
* Significant hematologic or hepatic abnormality
* Continuous requirement for supplemental oxygen
* Intercurrent infection at initiation of everolimus
* Embolization of angiomyolipoma within one month; any other recent surgery within 2 months of initiation of everolimus
* Pregnant or lactating women
* Use of an investigational drug within the last 30 days
* Must be adequately recovered from the acute toxicities of any prior therapy
* Clinical evidence of impending herniation or focal neurologic deficit related to the subject's astrocytoma
* Unwilling or unable to use highly effective contraception

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2007-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David N Franz, M.D., Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

REFERENCES:
- [Derived] Peters JM, Prohl A, Kapur K, Nath A, Scherrer B, Clancy S, Prabhu SP, Sahin M, Franz DN, Warfield SK, Krueger DA. Longitudinal Effects of Everolimus on White Matter Diffusion in Tuberous Sclerosis Complex. Pediatr Neurol. 2019 Jan;90:24-30. doi: 10.1016/j.pediatrneurol.2018.10.005. Epub 2018 Oct 18. PMID 30424962
- [Derived] Sparagana S, Franz DN, Krueger DA, Bissler JJ, Berkowitz N, Burock K, Kingswood JC. Pooled analysis of menstrual irregularities from three major clinical studies evaluating everolimus for the treatment of tuberous sclerosis complex. PLoS One. 2017 Oct 12;12(10):e0186235. doi: 10.1371/journal.pone.0186235. eCollection 2017. PMID 29023494
- [Derived] Franz DN, Agricola K, Mays M, Tudor C, Care MM, Holland-Bouley K, Berkowitz N, Miao S, Peyrard S, Krueger DA. Everolimus for subependymal giant cell astrocytoma: 5-year final analysis. Ann Neurol. 2015 Dec;78(6):929-38. doi: 10.1002/ana.24523. Epub 2015 Nov 9. PMID 26381530
- [Derived] Krueger DA, Care MM, Agricola K, Tudor C, Mays M, Franz DN. Everolimus long-term safety and efficacy in subependymal giant cell astrocytoma. Neurology. 2013 Feb 5;80(6):574-80. doi: 10.1212/WNL.0b013e3182815428. Epub 2013 Jan 16. PMID 23325902
- [Derived] Tillema JM, Leach JL, Krueger DA, Franz DN. Everolimus alters white matter diffusion in tuberous sclerosis complex. Neurology. 2012 Feb 21;78(8):526-31. doi: 10.1212/WNL.0b013e318247ca8d. Epub 2012 Jan 18. PMID 22262746
- [Derived] Krueger DA, Care MM, Holland K, Agricola K, Tudor C, Mangeshkar P, Wilson KA, Byars A, Sahmoud T, Franz DN. Everolimus for subependymal giant-cell astrocytomas in tuberous sclerosis. N Engl J Med. 2010 Nov 4;363(19):1801-11. doi: 10.1056/NEJMoa1001671. PMID 21047224

RESULTS

PARTICIPANT FLOW:
Groups:
- Everolimus: This was a non-randomized, open-label, single arm study; all patients in the study received treatment with everolimus.
Period: Overall Study
Arm/Group | Everolimus
Started | 28
Completed | 22
Not Completed | 6

BASELINE CHARACTERISTICS:
Arm/Group | Everolimus
Number analyzed (Participants) | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 22
  Between 18 and 65 years | 6
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 24
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 28

OUTCOME MEASURES:

1. Primary Outcome: Number With Observed Adverse Side Effects
Time Frame: During the entire study
Measure: Number; unit: participants
Groups:
- Everolimus: This was a non-randomized, open-label, single arm study; all patients in the study received treatment with everolimus. The initial starting dose was to be 3.0 mg/m2/day taken either daily or every other day with titration to achieve target trough concentrations of 5 to 15 ng/mL, subject to tolerability. Study drug was self-administered orally (or administered by a caregiver) at the same time each day.
Arm/Group | Everolimus
Number analyzed (Participants) | 28
participants
  Upper Respiratory Tract Infection | 26
  Stomatitis | 25
  Sinusitis | 15
  Mouth Ulceration | 14
  Cellulitis | 12
  Diarrhoea | 12
  Gastroenteritis | 12
  Otitis Media | 11
  Pyrexia | 10
  Vomiting | 10
  Acne | 9
  Convulsion | 9
  Nasopharyngitis | 9
  Rhinitis Allergic | 9
  Conjunctivitis | 8
  Pharyngitis | 8
  Rash | 8
  Constipation | 7
  Cough | 7
  Dermatitis Acneiform | 7
  Dermatitis Contact | 7
  Excoriation | 7
  Laceration | 7
  Nasal Congestion | 7
  Otitis Externa | 7
  Abnormal Behaviour | 6
  Body Tinea | 6
  Dry Skin | 6
  Pneumonia | 6
  Skin Infection | 6
  Urinary Tract Infection | 6

2. Secondary Outcome: Overall Reduction in SEGA Tumor Volume.
Time Frame: During the entire study
Measure: Number; unit: participants
Arm/Group | Everolimus
Number analyzed (Participants) | 26
participants
  # with reductions > 30% relative to baseline | 14
  # with reductions > 50% relative to baseline | 12

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout the course of the study, which was open for seven years.
Arm/Group | Everolimus
Serious Adverse Events (participants affected / at risk) | 9/28
Other Adverse Events (participants affected / at risk) | 28/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Everolimus (N=28)
Abscess Limb (Infections and infestations) | 2 (2)
Cellulitis (Infections and infestations) | 2 (2)
Convulsion (Nervous system disorders) | 2 (2)
Bronchitis Viral (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Post Lumbar Puncture Syndrome (Injury, poisoning and procedural complications) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Sudden Unexplained Death In Epilepsy (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Everolimus (N=28)
Upper Respiratory Tract Infection (Infections and infestations) | 26 (26)
Sinusitis (Infections and infestations) | 15 (15)
Cellulitis (Infections and infestations) | 12 (12)
Gastroenteritis (Infections and infestations) | 12 (12)
Otitis media (Infections and infestations) | 11 (11)
Nasopharyngitis (Infections and infestations) | 9 (9)
Pharyngitis (Infections and infestations) | 8 (8)
Otitis Externa (Infections and infestations) | 7 (7)
Pneumonia (Infections and infestations) | 6 (6)
Skin infection (Infections and infestations) | 6 (6)
Urinary Tract Infection (Infections and infestations) | 6 (6)
Stomatitis (Gastrointestinal disorders) | 25 (25)
Mouth Ulceration (Gastrointestinal disorders) | 14 (14)
Diarrhoea (Gastrointestinal disorders) | 6 (6)
Acne (Skin and subcutaneous tissue disorders) | 8 (8)
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 7 (7)
Pyrexia (General disorders) | 8 (8)
Conjunctivitis (Eye disorders) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes